CLINICAL TRIAL: NCT02328391
Title: MULTICENTER, PROSPECTIVE, OBSERVATIONAL OF ERLOTINIB AS SECOND-LINE TREATMENT IN PATIENTS WITH NON-SMALL CELL (NSCLC) LUNG CANCER WITH PREDOMINANTLY SQUAMOUS HISTOLOGY AND CARRIERS OF THE GENE (EGFR) EPIDERMAL GROWTH FACTOR RECEPTOR NATIVE
Brief Title: STUDY OBSERVATIONAL OF ERLOTINIB AS SECOND LINE TREATMENT IN PATIENTS WITH SQUAMOUS NSCLC AND EGFR NATIVE
Acronym: GGCP 055/12
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo Gallego de Cancer de Pulmon (Other)
Responsible Party: Sponsor
Other Study IDs: GGC-ERL-2012-01
Record Dates: First submitted 2014-04-24; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-09

CONDITIONS: Carcinoma, Squamous Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
OBJECTIVE study the effectiveness of the administration of Erlotinib 150 mg/Day v.o. in second-line treatment in patients with lung cancer advanced non-small of histology predominantly flaky by assessing the survival free of progression (SLP).

Design Studio postautoritation of multicenter observational follow-up prospective (EPA-SP) type.

DISEASE OTRASTORNO A study of cell Lung Cancer not small (NSCLC). MEDICATION object data to study the drug under study is erlotinib.

-Dose and treatment guidelines follow the corresponding product sheet. Management of dosage and adverse effects specified in point H. 15 of the Protocol.

POPULATION in study and number TOTAL of subjects population under study: adult patients with diagnosis of NSCLC with predominantly squamous histology total number of subjects: the participation of approximately 51 patients is expected DISEASE OR DISORDER TO STUDY Non Small Cell Lung Cancer (NSCLC). MEDICATION DATA OBJECT OF STUDY The drug under study is erlotinib.

-Dose and treatment guidelines Follow the corresponding product sheet. Management of dosage and adverse effects specified in point H. 15 of the Protocol.

STUDY POPULATION AND NUMBER TOTAL OF SUBJECTS Study: adult patients with diagnosis of NSCLC with predominantly squamous histology total number of subjects: the participation of approximately 51 patients is expected.

ELIGIBILITY:
Inclusion Criteria:

-• Age ≥ 18 years.

* Histological or cytologic diagnosis of cancer (NSCLC) with predominantly squamous histology stage IV non-small-cell lung.
* ECOG performance status between 0 and 2.
* Patients who have progressed to a first line of advanced disease and are eligible for a second line with Erlotinib.
* Patients that grant informed, preferably in writing, or oral consent before witnesses independent of the research team.

Exclusion Criteria:

-• Patients with uncontrolled or severe systemic disease, an active infection, neoplasia concomitant or secondary neoplasia to primary disease, except for carcinoma in situ of cervix or adequately treated skin carcinoma.

* Disease with mutated EGFR, according to local laboratory. The determination of the EGFR is not mandatory. Those patients from centers where there is the determination of the EGFR or those patients that the EGFR is unknown may be included in.
* Inability to take oral medication or previous surgical procedures that affect the absorption and imply the need for intravenous or parenteral feeding.
* Interstitial lung disease clinically active.
* Unstable angina or recent myocardial infarction.
* Brain metastasis uncontrolled and progressive.
* Patients who are participating in a clinical trial.
* Use of an inhibitor of tyrosine kinase in first line of treatment.
* Patients whose estimated life expectancy does not reach the 2 months.
* Any condition, situation which, in the opinion of the investigator, may endanger the safety of the patient, or could interfere significantly with the involvement of the subject in the study or evaluation of the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosis of NSCLC with predominantly squamous histology. The subject shall be considered included in the study when, fulfilling the criteria of selection, accept their participation therein by the signing of informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-03 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Study the effectiveness of the administration of Erlotinib in 2nd line treatment in patients with advanced NSCLC scaly through assessment of the SLP | Collect the available information of the visits made by the patient according to the usual practice up to a max of 9 m after the inclusion of the last patient.

SECONDARY OUTCOMES:
Determination TR y TCE. • Determinar SG. • Identificar los diferentes factores pronósticos relacionados con la SLP y SG. • Determinar el perfil de seguridad del tratamiento. | Collect the available information of the visits made by the patient according to the usual practice up to a max of 9 m after the inclusion of the last patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Gallego Cancer de Pulmon, Santiago de Compostela, A Coruña, Spain